CLINICAL TRIAL: NCT07343180
Title: The Effect of Acceptance and Commitment Therapy-Based Psychoeducation on Self-Esteem and Interpersonal Problem-Solving Skills in Youth With Social Media Addiction
Brief Title: ACT-Based Psychoeducation for Youth With Social Media Addiction
Acronym: ACT-SM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Kahramanmaras Sutcu Imam University (Other)
Collaborators: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Zeynep KEKEÇ, Research Assistant, Department of Psychiatric Nursing, Kahramanmaras Sutcu Imam University, Kahramanmaras Sutcu Imam University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: KSU-TAREK-2025/15-04
Record Dates: First submitted 2025-12-01; First posted 2026-01-15 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2025-12

CONDITIONS: Social Media Addiction; Self Esteem; Interpersonal Problem; Problem-solving
Keywords: Social Media Addiction; Acceptance and Commitment Therapy (ACT); Psychoeducation; Interpersonal Problem-Solving; Self-Esteem; Behavioral Addiction
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either the intervention group, which will receive an 8-session ACT-based psychoeducational program, or the control group, which will not receive any intervention during the study period. Randomization will be performed using Research Randomizer by a statistician not involved in the study. The intervention and control groups will each consist of 37 participants. Both groups will complete assessments at baseline (pre-test), interim follow-up, and post-test using validated scales for self-esteem, interpersonal problem-solving skills, and social media addiction. The control group will receive a single psychoeducation session after the follow-up assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group - ACT-Based Psychoeducation (Experimental): Participants in this group will receive an 8-session Acceptance and Commitment Therapy (ACT)-based psychoeducational program designed to improve self-esteem and interpersonal problem-solving skills while reducing social media addiction. Assessments will be conducted at baseline (pre-test), interim follow-up, and post-test, using validated scales. The intervention will be delivered in groups of 37 participants by a trained researcher.
  Interventions: Behavioral: ACT-Based Psychoeducational Program
- Control Group - No Intervention (Waitlist) (No Intervention): Participants in this group will not receive any intervention during the study period. Assessments will be conducted at the same time points as the intervention group (baseline, interim follow-up, and post-test) using the same validated scales. After the 2-month follow-up, participants will receive a single psychoeducation session.

INTERVENTIONS:
Behavioral: ACT-Based Psychoeducational Program — The intervention consists of an 8-session Acceptance and Commitment Therapy (ACT)-based psychoeducational program aimed at improving self-esteem and interpersonal problem-solving skills and reducing social media addiction among young adults. Sessions will be delivered in small groups of 6-7 participants by a trained researcher with certification in ACT and psychoeducation.
  Assessments will be conducted at three time points: baseline (pre-test), interim follow-up, and post-test. During the program, participants will engage in ACT exercises, mindfulness practices, and value-based activities, focusing on psychological flexibility, coping with negative internal experiences, and enhancing effective interpersonal strategies.
  Participants will also complete validated scales for self-esteem, interpersonal problem-solving, and social media addiction at each assessment point.
  Arms: Intervention Group - ACT-Based Psychoeducation

SUMMARY:
While social media offers opportunities for connection and self-expression, it also brings significant challenges, particularly social media addiction, characterized by excessive and uncontrolled use. Although not officially recognized as a diagnostic category, its inclusion among behavioral addictions reflects its growing impact on mental health. Social media addiction may lead to psychological symptoms such as family and social conflicts, stress due to unmet responsibilities, anxiety, and irritability. This problem has become especially critical among young people. A 2025 meta-analysis found the prevalence of social media addiction among university students to be 18.4% and reported negative effects on academic achievement. Research also shows that social media addiction is associated with decreased self-esteem, emotion regulation difficulties, and dysfunctional interpersonal relationships. Social comparison tendencies and idealized digital identity presentations further harm young individuals' self-perceptions, contributing to low self-esteem and social anxiety.

Interpersonal difficulties experienced in relationships are defined as "interpersonal problems," while the cognitive-behavioral processes used to resolve these difficulties are called "interpersonal problem solving." These skills are essential for effective conflict resolution, social adaptation, relationship quality, and overall well-being. Social media shapes both the emergence and resolution of interpersonal problems; however, current knowledge in this area is limited. Excessive use contributes to interpersonal conflicts, deterioration of relationships, and reduced face-to-face communication. Thus, social media addiction may impair interpersonal problem-solving skills by disrupting daily functioning.

Although the literature includes correlational studies on social media addiction, self-esteem, and interpersonal functioning, research testing Acceptance and Commitment Therapy (ACT)-based psychoeducation remains scarce. This study offers a theoretical contribution by applying a third-wave therapy approach to the psychosocial challenges of the digital age. It aims to evaluate the effects of an ACT-based psychoeducation program developed for young individuals with social media addiction on self-esteem and interpersonal problem-solving skills. Given the limited number of such programs in Türkiye, this study is original and aims to fill an important gap in the literature.

DETAILED DESCRIPTION:
The widespread use of technology and early access to digital devices have significantly increased in recent years. Continuous connectivity, mobility, and affordability allow users to interact freely with social media. Young individuals often integrate mobile devices into daily routines, spend excessive time online, and keep devices nearby even during sleep. While social media allows relationship-building and self-expression, excessive and uncontrolled use may lead to social media addiction. Although not officially recognized in psychiatric diagnostic systems, its classification under behavioral addictions reflects its increasing impact on mental health. Behavioral addictions may cause family and social conflicts, stress due to unmet responsibilities, anxiety, and irritability.

Social media addiction is particularly prevalent among young adults. A 2025 meta-analysis reported a prevalence rate of 18.4% among university students and its negative effects on academic performance. Another study with 1,215 students found higher addiction levels associated with increased depression scores. Excessive use also affects body dissatisfaction and self-esteem. These findings show that social media addiction decreases self-esteem, disrupts emotional regulation, and impairs interpersonal functioning. Social comparison tendencies and idealized digital identities may worsen self-perceptions, contributing to low self-esteem and social anxiety.

Multiple studies have shown significant negative relationships between social media addiction and self-esteem. Facebook addiction has been linked to low self-esteem. Similarly, low self-esteem was associated with higher social media addiction scores. Research from Ecuador reported moderate negative effects of social media addiction on self-esteem and well-being. A 2023 adolescent study found that addiction negatively predicted self-esteem and body image. Self-esteem is a fundamental construct related to life satisfaction, self-efficacy, psychological resilience, and interpersonal relationships.

Interpersonal difficulties are defined as "interpersonal problems," while cognitive and behavioral processes intended to reduce tension in these areas are conceptualized as "interpersonal problem-solving." Interpersonal problem-solving skills enable constructive conflict resolution and support social adaptation, relationship quality, and well-being. Social media influences how individuals generate and solve interpersonal problems, though evidence is limited. Excessive use leads to relationship deterioration, communication restrictions, and increased interpersonal conflicts. Social media addiction may impair interpersonal problem-solving due to its negative impact on overall functioning. Additionally, individuals with higher interpersonal problem-solving skills show lower addiction levels. Internet addiction has also been associated with avoidance-oriented coping.

Acceptance and Commitment Therapy (ACT), a mindfulness-based intervention focusing on psychological flexibility, encourages individuals to accept internal experiences and act in accordance with personal values. ACT promotes awareness of thoughts and emotions and engagement in value-driven behaviors. Research demonstrates its effectiveness for anxiety, depression, addictive behaviors, and self-perception. ACT-based interventions have reduced social media use and decreased psychological distress in university students. ACT has also been found effective in reducing FOMO and increasing psychological flexibility.

ACT has improved self-esteem and interpersonal problem-solving in diverse populations, such as individuals with schizophrenia, PCOS, body dysmorphic disorder, and obesity. ACT reduced internet addiction components and interpersonal difficulties among high school students. It also improved adolescents' interpersonal skills and was comparable to CBT in addressing interpersonal problems.

Despite the correlational evidence linking social media addiction to self-esteem and interpersonal functioning, ACT-based interventions remain limited, especially for young adults. Thus, our study offers theoretical and practical innovation by applying a third-wave therapy model to digital-age psychosocial problems. The study aims not only to reduce addictive behaviors but also to improve psychological flexibility, self-esteem, and interpersonal problem-solving skills. Findings are expected to guide mental health professionals, psychiatric nurses, counselors, and university guidance services.

The study also aligns with the 12th Development Plan (2024-2028), which emphasizes informing youth about digital risks, supporting evidence-based policy design, and promoting healthy technology use.

Hypotheses H1a: ACT-based psychoeducation increases self-esteem. H1b: ACT-based psychoeducation reduces ineffective interpersonal problem-solving.

H1c: ACT-based psychoeducation enhances effective interpersonal problem-solving.

H1d: ACT-based psychoeducation reduces social media addiction.

Study Design This randomized controlled trial (RCT) will be conducted at Kahramanmaraş Sütçü İmam University between November 1, 2025, and September 30, 2026. A 2×3 split-plot design (intervention/control × pretest/posttest/follow-up) will be used. Assessments will occur at baseline, post-intervention, and two-month follow-up.

Study Population and Sample The study population includes students aged 18-30 enrolled between 01/05/2025 and 01/06/2026. Based on GPower calculations (effect size d = 0.30; α = .05; power = .90), 31 participants per group were required. With 20% added for attrition, the total sample is 74 (37 per group). Intervention groups will consist of approximately 7-8 participants.

Randomization Participants scoring ≥4 on the SMAS-AF will be randomized using simple randomization (Research Randomizer). A statistician not involved in the study will manage allocation.

Variables Independent variable: ACT-based psychoeducation program

Dependent variables:

Rosenberg Self-Esteem Scale (RSES) Social Media Addiction Scale-Adult Form (SMAS-AF) Interpersonal Problem-Solving Inventory

Data Collection Tools Information Form; Rosenberg Self-Esteem Scale (RSES); Social Media Addiction Scale-Adult Form (SMAS-AF); Interpersonal Problem-Solving Inventory.

Implementation Baseline assessments will be completed face-to-face. The intervention group will attend eight ACT-based psychoeducation sessions administered by psychiatric nurse Zeynep Kekeç, certified in psychoeducation and ACT. Post-test assessments will be completed in the final session. The control group will not receive intervention during the study but will be offered a one-session program afterward.

Data Analysis Data will be analyzed in SPSS. Normality will be assessed using the Shapiro-Wilk test. Descriptive statistics will be calculated. Parametric or non-parametric analyses will be selected based on distribution. Cronbach's alpha values will be computed. Significance level: p < 0.05.

Ethical Considerations Ethical approval was obtained from the Kahramanmaraş Sütçü İmam University Medical Research Ethics Committee. Permissions for scales were secured. Participation is voluntary, and confidentiality and withdrawal rights will be ensured.

ELIGIBILITY:
Inclusion Criteria:

* Voluntary participation in the study.
* Age between 18 and 30 years.
* Social Media Addiction Scale - Adult Form (SMAS-AF) item average score of 4 or higher.

Exclusion Criteria:

* Hearing or speech impairments that would prevent completing the surveys.
* Currently participating in a similar psychoeducational program.
* Receiving treatment for any psychiatric disorder at the time of the study.

Withdrawal Criteria:

* Missing two consecutive sessions
* Disruptive behavior
* Non-compliance with group rules
* Failure to complete session assignments

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 74 (Estimated)
Dates: Start 2026-01-10 (Estimated); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Social Media Addiction - Social Media Addiction Scale - Adult Form (SMAS-AF) | Baseline (Pre-test), Interim Follow-up (at the end of the 8-week intervention), Post-test (8 weeks after the "interim follow-up")
  ACT-based psychoeducational intervention reduces participants' levels of social media addiction. The SMAS-AF comprises 20 items across two sub-dimensions: "Virtual Tolerance" and "Virtual Communication". The total score that can be obtained from the scale varies between 20 and 100, with higher scores indicating higher levels of social media addiction.
Self-Esteem - Rosenberg Self-Esteem Scale (RSES) | Baseline (Pre-test), Interim Follow-up (at the end of the 8-week intervention), Post-test (8 weeks after the "interim follow-up")
  ACT-based psychoeducational intervention increases participants' levels of self-esteem. Total scores range from 0 to 6, with 0-1 indicating high self-esteem, 2-4 moderate self-esteem, and 5-6 low self-esteem.
Interpersonal Problem-Solving Skills | Baseline (Pre-test), Interim Follow-up (at the end of the 8-week intervention), Post-test (8 weeks after the "interim follow-up")
  ACT-based psychoeducational intervention increase participants' ability to solve interpersonal problems. The instrument which is a five-point lichert scale comprised five sub-scales and 50 items in total. The items range from 1 (Completely inappropriate) to 5 (Completely appropriate). The high score received for each sub-scale indicates that the quality of solving interpersonal problem is also high. The five sub-scales are; negative approach to the problem (NA), constructive problem solving (CPS), lack of self-confidence (LSC), Irresponsiveness (I), and persistent-steadfast approach (PA). The number of items included in each subscale is respectively; 16, 16, 7, 5, and 6.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep KEKEÇ, PhD student, Study Chair — Kahramanmaraş Sütçü İmam University, Faculty of Health Sciences; Döndü ÇUHADAR, PhD, Study Director — Gaziantep University, Faculty of Health Sciences
Locations (1):
- Kahramanmaraş Sütçü İmam Üniversitesi, Faculty of Health Sciences, Kahramanmaraş, Onikişubat, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data from this study will not be shared to protect participant privacy and confidentiality. The data contain sensitive information regarding mental health and social media use of young adults, and sharing de-identified data could still pose a risk of re-identification. The study team will use the data exclusively for the purposes of the current research and related publications.

REFERENCES:
- [Background] Masoumian S, Ashouri A, Ghomian S, Keshtkar M, Siahkamary E, Vahed N. Efficacy of Acceptance and Commitment Therapy Compared to Cognitive Behavioral Therapy on Anger and Interpersonal Relationships of Male Students. Iran J Psychiatry. 2021 Jan;16(1):21-29. doi: 10.18502/ijps.v16i1.5374. PMID 34054979
- [Background] Bernal-Manrique, K. N., García-Martín, M. B., ve Ruiz, F. J. 2020. "Effect of acceptance and commitment therapy in improving interpersonal skills in adolescents: A randomized waitlist control trial", Journal of Contextual Behavioral Science, 17, 86-94.
- [Background] Firouzkouhi Berenjabadi, M., Pourhosein, M., ve Ghasemi Argene, M. 2021. "The effectiveness of acceptance and commitment therapy (ACT) on interpersonal difficulties and internet addiction among high school students", Journal of Applied Psychological Research, 12(2), 283-301. https://doi.org/10.22059/japr.2021.310151.643639
- [Background] Alavi Hajazi, F., ve Nezhadmohammad Nameghi, A. 2018. "The effect of group training based on acceptance and commitment on reducing anxiety and interpersonal problems in obese women", Journal of Research in Health, 8(6), 522-530.http://jrh.gmu.ac.ir/article-1-1481-en.html
- [Background] Dehbaneh, M. A. 2019. "Effectiveness of acceptance and commitment therapy in improving interpersonal problems, quality of life, and worry in patients with body dysmorphic disorder". Electronic Journal of General Medicine, 16(1).
- [Background] Shi JY, Cao YM, Luo HY, Liu S, Yang FM, Wang ZH. Effect of a group-based acceptance and commitment therapy (ACT) intervention on self-esteem and psychological flexibility in patients with schizophrenia in remission. Schizophr Res. 2023 May;255:213-221. doi: 10.1016/j.schres.2023.03.042. Epub 2023 Apr 1. PMID 37012184
- [Background] Moradi F, Ghadiri-Anari A, Dehghani A, Reza Vaziri S, Enjezab B. The effectiveness of counseling based on acceptance and commitment therapy on body image and self-esteem in polycystic ovary syndrome: An RCT. Int J Reprod Biomed. 2020 Apr 30;18(4):243-252. doi: 10.18502/ijrm.v13i4.6887. eCollection 2020 Apr. PMID 32494763
- [Background] Bal, P. N., Kahraman, S., Hündür, U. 2025. "A correlational study of social media-related FoMO and psychological flexibility among adults: An acceptance and commitment therapy perspective". Asia Pacific Journal of Counselling and Psychotherapy. Advance online publication. https://doi.org/10.1080/21507686.2025.2495147
- [Background] Marmer, L. W., Nurwianti, F. 2020. "Group acceptance and commitment therapy to reduce psychological distress among college students with social media addiction". Proceedings of the 3rd International Conference on Intervention and Applied Psychology (ICIAP 2019) and the 4th Universitas Indonesia Psychology Symposium for Undergraduate Research (UIPSUR 2019), 132-143. Atlantis Press. https://doi.org/10.2991/assehr.k.201125.011
- [Background] Gloster, A. T., Walder, N., Levin, M. E., Twohig, M. P., Karekla, M. 2020. "The empirical status of acceptance and commitment therapy: A review of meta-analyses". Journal of Contextual Behavioral Science, 18, 181-192
- [Background] Twohig MP, Levin ME. Acceptance and Commitment Therapy as a Treatment for Anxiety and Depression: A Review. Psychiatr Clin North Am. 2017 Dec;40(4):751-770. doi: 10.1016/j.psc.2017.08.009. PMID 29080598
- [Background] Hayes SC, Luoma JB, Bond FW, Masuda A, Lillis J. Acceptance and commitment therapy: model, processes and outcomes. Behav Res Ther. 2006 Jan;44(1):1-25. doi: 10.1016/j.brat.2005.06.006. PMID 16300724
- [Background] Hayes, S. C., Strosahl, K. D., Wilson, K. G. 1999. Acceptance and commitment therapy: An experiential approach to behavior change. New York: Guilford Press.
- [Background] Ahmad, S., Nurwianti, F. 2020. "Using Acceptance and Commitment Therapy (ACT) in a group setting to increase quality of life in university students with social media addictions". Proceedings of the 2nd Tarumanagara International Conference on the Applications of Social Sciences and Humanities (TICASH 2020). Atlantis Press. https://doi.org/10.2991/assehr.k.201125.015
- [Background] Hasan AA, Jaber AA. Prevalence of internet addiction, its association with psychological distress, coping strategies among undergraduate students. Nurse Educ Today. 2019 Oct;81:78-82. doi: 10.1016/j.nedt.2019.07.004. Epub 2019 Jul 12. PMID 31352247
- [Background] Berezovskaya, I. P., Shipunova, O. D., Kedich, S. I. 2019. "Internet addiction and youth coping strategies". Proceedings of the XI International Scientific Conference on Communicative Strategies of the Information Society, 1-6. Atlantis Press.
- [Background] Şahin, S., İbili, E., Uluyol, Ç. 2017. "Öğretmen adaylarında problem çözme eğilimi ve internet bağımlılığı ilişkisinin incelenmesi", Afyon Kocatepe University Journal of Social Sciences, 19(1), 1-21.
- [Background] Mercan N, Uysal B. The relationship of social media addiction with interpersonal problem-solving and personality traits in university students. Arch Psychiatr Nurs. 2023 Apr;43:50-56. doi: 10.1016/j.apnu.2022.12.025. Epub 2023 Jan 4. PMID 37032015
- [Background] İbili, E. 2017. "Internet addiction levels and problem-solving skills in the teaching profession: An investigation", Acta Didactica Napocensia, 10(4), 93-107.
- [Background] Yayman, E., Bilgin, O. 2020. "Relationship between social media addiction, game addiction and family functions", International Journal of Evaluation and Research in Education, 9(4), 979-986.
- [Background] Jiang, F., Lu, S., Zhu, X., Song, X. 2021. "Social media impacts the relation between interpersonal conflict and job performance", Asia Pacific Journal of Human Resources, 59(3), 420-441.
- [Background] Çam, S., Tümkaya, S. 2007. "Developing the interpersonal problem-solving inventory (IPSI): The validity and reliability process", Turkish Psychological Counseling and Guidance Journal, 3(28), 95-111.
- [Background] Orth, U., Robins, R. W. 2014. "The development of self-esteem", Current Directions in Psychological Science, 23(5), 381-387.
- [Background] Rosenberg, M. 1965. Society and the adolescent self-image. Princeton: Princeton University Press.
- [Background] Colak M, Bingol OS, Dayi A. Self-esteem and social media addiction level in adolescents: The mediating role of body image. Indian J Psychiatry. 2023 May;65(5):595-600. doi: 10.4103/indianjpsychiatry.indianjpsychiatry_306_22. Epub 2023 May 15. PMID 37397839
- [Background] Oleas Rodríguez, D., ve López-Barranco Pardo, G. 2024. "The impact of social media addiction on state self-esteem; a cross-sectional study in university students from Samborondón, Ecuador", European Public & Social Innovation Review, 9, 1-15. https://doi.org/10.31637/epsir-2024-1042
- [Background] Andreassen CS, Pallesen S, Griffiths MD. The relationship between addictive use of social media, narcissism, and self-esteem: Findings from a large national survey. Addict Behav. 2017 Jan;64:287-293. doi: 10.1016/j.addbeh.2016.03.006. Epub 2016 Mar 19. PMID 27072491
- [Background] Vogel, E. A., Rose, J. P., Roberts, L. R., ve Eckles, K. 2014. "Social comparison, social media, and self-esteem", Psychology of Popular Media Culture, 3(4), 206-222.
- [Background] Hawi, N. S., ve Samaha, M. 2017. "The relations among social media addiction, self-esteem, and life satisfaction in university students", Social Science Computer Review, 35(5), 576-586
- [Background] Błachnio, A., Przepiorka, A., ve Pantic, I. 2016. "Association between Facebook addiction, self-esteem and life satisfaction", Computers in Human Behavior, 55, 701-705.
- [Background] Khan, M. A., Alvi, S. M., Hafeez, S., Akhtar, S., ve Younis, K. 2025. "The impact of media exposure on self-esteem and body-satisfaction among youth: The moderating role of resilience", ACADEMIA International Journal for Social Sciences, 4(2), 2237-2252.
- [Background] Salari N, Zarei H, Rasoulpoor S, Ghasemi H, Hosseinian-Far A, Mohammadi M. The impact of social networking addiction on the academic achievement of university students globally: A meta-analysis. Public Health Pract (Oxf). 2025 Jan 13;9:100584. doi: 10.1016/j.puhip.2025.100584. eCollection 2025 Jun. PMID 39896338
- [Background] Woods HC, Scott H. #Sleepyteens: Social media use in adolescence is associated with poor sleep quality, anxiety, depression and low self-esteem. J Adolesc. 2016 Aug;51:41-9. doi: 10.1016/j.adolescence.2016.05.008. Epub 2016 Jun 10. PMID 27294324
- [Background] Nakayama H, Ueno F, Mihara S, Kitayuguchi T, Higuchi S. Relationship between problematic Internet use and age at initial weekly Internet use. J Behav Addict. 2020 Apr 1;9(1):129-139. doi: 10.1556/2006.2020.00009. PMID 32359236
- [Background] Cheng C, Lau YC, Chan L, Luk JW. Prevalence of social media addiction across 32 nations: Meta-analysis with subgroup analysis of classification schemes and cultural values. Addict Behav. 2021 Jun;117:106845. doi: 10.1016/j.addbeh.2021.106845. Epub 2021 Jan 26. PMID 33550200
- [Background] Çiftçi, H. 2018. "Social media addiction in university students", MANAS Journal of Social Studies, 7(4), 417-434.
- [Background] Hruska, J., ve Maresova, P. 2020. "Use of social media platforms among adults in the United States-Behavior on social media", Societies, 10(1), 27. https://doi.org/10.3390/soc10010027
- [Background] Kabali HK, Irigoyen MM, Nunez-Davis R, Budacki JG, Mohanty SH, Leister KP, Bonner RL Jr. Exposure and Use of Mobile Media Devices by Young Children. Pediatrics. 2015 Dec;136(6):1044-50. doi: 10.1542/peds.2015-2151. Epub 2015 Nov 2. PMID 26527548
- [Background] Bülbül, H., ve Tunç, T. 2018. "Phone and game addiction: Scale analysis, the starting age and its relationship with academic success", Süleyman Demirel University Visionary Journal, 9(21), 1-13. https://doi.org/10.21076/vizyoner.431446
- See also: Presidency of the Republic of Turkey, Presidency of Strategy and Budget. 2023. "Twelfth Development Plan (2024-2028)." — https://www.sbb.gov.tr/wp-content/uploads/2023/12/On-Ikinci-Kalkinma-Plani_2024-2028_11122023.pdf
- See also: Republic of Turkey Ministry of Health. (2018). National Strategy Document and Action Plan for Combating Behavioral Addictions (2019-2023). Directorate of Communications of the Republic of Turkey. — https://imyo.deu.edu.tr/wp-content/uploads/2021/12/davranissal-bagimliliklar-ile-mucadele-ulusal-strateji-belgesi-ve-eylem-plani-2018-2023pdf_compressed.pdf

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan: Study Protocol and Statistical Analysis Plan (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT07343180/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-07): https://cdn.clinicaltrials.gov/large-docs/80/NCT07343180/ICF_001.pdf